CLINICAL TRIAL: NCT03665610
Title: A Phase 1, Multi-center, Extension Study to Further Evaluate the Safety, Pharmacodynamics and Pharmacokinetics of Ozanimod and Active Metabolites in Healthy Adult Subjects
Brief Title: Extension Study to Further Evaluate the Safety, Pharmacodynamics and Pharmacokinetics of Ozanimod and Active Metabolites
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: RPC01-1915; U1111-1219-5905 (Registry Identifier: WHO)
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacodynamics; Pharmacokinetics; Ozanimod; Safety; Healthy Subjects
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mandatory Safety Population: All subjects who enrolled in studies RPC01-1912, RPC01-1913, or RPC01-1914 and received at least one dose of ozanimod or IP (per parent studies), excluding subjects who discontinued during Period 1 of study RPC01-1913.
  Interventions: Drug: ozanimod
- Optional pharmacokinetic(s) and pharmacodynamics(s) population: Subjects in study RPC01-1913 have completed the study at least through Period 2 and completed the 7 ± 2 days postdose follow-up assessments; or subjects in study RPC01-1914 have completed the study through the 7 ± 2 days postdose follow-up and had no major protocol violations in the parent studies that are deemed to impact PK or PD assessments.

INTERVENTIONS:
Drug: ozanimod — ozanimod
  Groups: Mandatory Safety Population

SUMMARY:
Study Design

This is a Phase 1, multi-center, extension study to collect safety data up to 75 ± 10 days postdose from the Phase 1 studies RPC01-1912, RPC01-1913 and RPC01-1914 (ie, the "parent studies") and PK/PD data up to 75 ± 10 days postdose from studies RPC01-1913 and RPC01-1914. This study consists of two parts:

* Mandatory data collection for safety: Subjects enrolled in the parent studies were consented to have data on adverse events (AEs), serious adverse events (SAEs), pregnancy test results, and concomitant medications up to the 75 ± 10 days postdose follow-up collected and reported in this study.
* Optional sparse sampling for PK/PD: Eligible subjects from studies RPC01-1913 and RPC01-1914 will be offered the opportunity to return to the clinical research unit (CRU) at four separate occasions for PK/PD sample collections up to the 75 ± 10 days postdose follow-up. After signing the informed consent form, eligible subjects will be randomized to one of three sequences with stratification by site/protocol. Subjects will return to the CRU in the morning (between approximately 8 am and 11 am) once at each of the four time windows.

Study Population The approximate number of subjects will be 230 for safety data and 129 for PK/PD data.

Length of Study The study duration is up to 84 days.

ELIGIBILITY:
Inclusion Criteria:

1. For the mandatory data collection for safety, subjects who enrolled in the Phase 1 studies RPC01-1912, RPC01-1913, or RPC01-1914 and received at least one dose of ozanimod or investigational product (IP) as applicable per the parent studies are eligible, except for subjects who discontinued during Period 1 of study RPC01-1913.
2. For the optional sparse sampling for PK/PD, subjects must satisfy the following criteria:

   1. Subjects in study RPC01-1913 have completed the study at least through Period 2 and completed the 7 ± 2 days postdose follow-up assessments; or subjects in study RPC01-1914 have completed the study through the 7 ± 2 days postdose follow-up.
   2. Subjects had no major protocol violations in the parent studies that are deemed to impact PK or PD assessments.
   3. Subjects must be able to comprehend and provide written informed consent, and must be able to comply with the requirements of the study, including the study visit schedule and other protocol requirements or restrictions.

Exclusion Criteria:

No Exclusion Criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The approximate number of subjects will be 230 for safety data (from parent studies RPC01-1912, RPC01-1913, and RPC01-1914) and 129 for PK/PD data (from parent studies RPC01-1913 and RPC01-1914).
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | From enrollment up to 75 +/- 10 days after the last dose in the parent study (RPC01-1912, RPC01-1913, or RPC01-1914)
  The incidence, severity, and relationship of TEAEs.

SECONDARY OUTCOMES:
Pharmacodynamics - absolute lymphocyte count (ALC) | Up to 75 +/- 10 days after the last dose in the parent study (RPC01-1913 or RPC01-1914)
  The absolute lymphocyte count (ALC) will be determined via hematology test
Pharmacodynamics - lymphocyte subsets | Up to 75 +/- 10 days after the last dose in the parent study (RPC01-1913 or RPC01-1914)
  Lymphocyte subsets will be measured using the immune cell monitoring epigenetic platform

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene
Locations (2):
- United States (2):
  - PPD Phase 1 Clinic, Austin, Texas
  - ICON Early Phase Services, LLC, San Antonio, Texas